CLINICAL TRIAL: NCT06033963
Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Carotid Artery Stenosis Undergoing Carotid EndArterectomy: A Pilot, Randomized Controlled Trial
Brief Title: Safety and Efficacy of Remote Ischemic Conditioning in Patients With Carotid Artery Stenosis Undergoing Carotid EndArterectomy
Acronym: SERIC-CASCEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERIC-CASCEA
Record Dates: First submitted 2023-09-03; First posted 2023-09-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carotid Artery Stenosis
Keywords: Remote ischemic conditioning; Carotid artery stenosis; Carotid endarterectomy
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC+CEA+Standard medical treatment (Active Comparator): Remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mmHg. RIC will be conducted twice daily for 6 consecutive days after enrollment. Additionally, the patients will be treated with carotid endarterectomy (CEA) and standard medical treatment according to the Chinese guideline for the secondary prevention of ischemic stroke and transient ischemic attack 2022.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC+CEA+Standard medical treatment (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mmHg. RIC will be conducted twice daily for 6 consecutive days after enrollment. Additionally, the patients will be treated with carotid endarterectomy (CEA) and standard medical treatment according to the Chinese guideline for the secondary prevention of ischemic stroke and transient ischemic attack 2022.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 200 mmHg.
  Arms: RIC+CEA+Standard medical treatment
Procedure: Sham remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 5 cycles of 5 min of bilateral upper limbs ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflations of a blood pressure cuff to 60 mmHg.
  Arms: Sham RIC+CEA+Standard medical treatment

SUMMARY:
The purpose of this study is to explore the safety and efficacy of remote ischemic conditioning in patients with carotid artery stenosis undergoing carotid endarterectomy.

DETAILED DESCRIPTION:
In this study, 100 patients with carotid artery stenosis undergoing carotid endarterectomy are included in our center in China according to the principle of random, and parallel control. The experimental group receive basic treatment and remote ischemic conditioning for 200mmHg, 2 times per day for 6 consecutive days. The control group receive basic treatment and remote ischemic conditioning control for 60mmHg, 2 times per day for 6 consecutive days. Two groups will be followed up for 1 year to evaluate the safety and efficacy of remote ischemic conditioning in patients with carotid artery stenosis undergoing carotid endarterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years, <80 years, regardless of sex;
2. Symptomatic or asymptomatic carotid artery stenosis. In symptomatic patients the degree of stenosis should more than 50% (Based on North American Symptomatic Carotid Endarterectomy Trial Collaborators (NASCET) Criteria), in asymptomatic patients the degree of stenosis should more than 70% (Based on NASCET Criteria);
3. Baseline mRS 0-2;
4. Can cooperate with and complete brain magnetic resonance imaging (MRI) examination;
5. Signed and dated informed consent is obtained;

Exclusion Criteria:

1. Evolving stroke;
2. Chronic complete occlusion of the carotid artery without obvious symptoms of cerebral ischemia;
3. Severe dementia;
4. The causes of cardiogenic embolism, such as rheumatic mitral or aortic valve stenosis, artificial heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, left ventricular wall thrombosis or valve tumor, congestive heart failure, bacterial endocarditis, etc;
5. Uncontrolled hypertension (defined as systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg, despite medication taken at enrollment);
6. Severe hepatic and renal dysfunction (defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥3 times higher than the upper limit of the normal range, creatinine >265umol/l (3mg/dl));
7. The patients who have the contraindication of remote ischemic conditioning treatment, such as severe soft tissue injury, fracture or vascular injury in the upper limb. Acute or subacute venous thrombosis, arterial occlusive disease, subclavian steal syndrome, etc;
8. Pregnant or lactating women;
9. He/She is participating in other clinical research or has participated in other clinical research or has participated in this study within 3 months prior to admission;
10. Other conditions that the researchers think are not suitable for the group.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who got ≥1 new Diffusion Weighted Imaging (DWI)-positive lesions on post-treatment magnetic resonance imaging (MRI) Scans. | 6 days
  Patients underwent magnetic resonance imaging (including DWI)at baseline and 6 days after randomization.

SECONDARY OUTCOMES:
The number of new Diffusion Weighted Imaging (DWI)-positive lesions on post-treatment magnetic resonance imaging (MRI) Scans. | 6 days
  Patients underwent magnetic resonance imaging (including DWI)at baseline and 6 days after randomization.
The volume of new Diffusion Weighted Imaging (DWI)-positive lesions on post-treatment magnetic resonance imaging (MRI) Scans. | 6 days
  Patients underwent magnetic resonance imaging(including DWI) at baseline and 6 days after randomization.
Number of patients with cerebrovascular events, cardiovascular events or death. | 1 year
  Cerebrovascular events included ischemic stroke, transient ischemic attack (TIA), cerebral hemorrhage. Cardiovascular events included angina and myocardial infarction. Death included any reason caused death.
Proportion of patients with any side effects of Remote ischemic conditioning (RIC) treatment. | 6 days
  The side effects referred to any side effects of RIC or sham RIC treatment, not including the sides effect of medications and Carotid Endarterectomy (CEA).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD, PhD, Study Chair — Neuroscience Center, Department of Neurology, The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China